CLINICAL TRIAL: NCT02424214
Title: Artificial Oocyte Activation Comparing Tow Different Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Al Baraka Fertility Hospital (Other); Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IbnSina Oocyte activation
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Oocyte Fertilization
MeSH Terms: interventions — strontium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ca Ionophore group (Experimental): Artificial Oocyte activation with Ca Ionophore for 20 min after Intracytoplasmic Sperm Injection
  Interventions: Other: Artificial Oocyte activation; Drug: Ca Ionophore
- Strontium Chloride group (Experimental): Artificial Oocyte activation with Strontium Chloride for 60 min after Intracytoplasmic Sperm Injection
  Interventions: Other: Artificial Oocyte activation; Drug: Strontium Chloride
- Only Intracytoplasmic Sperm Injection (No Intervention): after Intracytoplasmic Sperm Injection Oocytes will cultured and incubated

INTERVENTIONS:
Other: Artificial Oocyte activation
  Arms: Ca Ionophore group; Strontium Chloride group
Drug: Ca Ionophore
  Arms: Ca Ionophore group
Drug: Strontium Chloride
  Arms: Strontium Chloride group

SUMMARY:
Comparing the efficacy of tow factors for artificial Oocyte Activation for poor quality Oocytes and Teratozoospermia patients.

DETAILED DESCRIPTION:
The IVF outcome had been varied widely with a good portion of total fertilization failure even after the most advanced procedure for this group of patient Intracytoplasmic Sperm Injection, many factors that had been tested for assisting the failed group of patient to be fertilized artificially like Ca Ionophore, Strontium Chloride and others but we decide to compare the clinically proven factors for the efficacy and safety in a well randomized clinical trial and monitor the embryogenesis and pregnancy within the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* previous fertilization failure
* poor quality Oocytes
* poor sperms

Exclusion Criteria:

* normal patients

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate ( % ) | 9 months

SECONDARY OUTCOMES:
Blastocyst rate ( % ) | 9 months

CONTACTS AND LOCATIONS:
Locations (3):
- Al Barka fertility center, Manama, Bahrain
- Egypt (2):
  - Banon Fertility Center, Asyut
  - Ibnsina IVF center, Sohag

REFERENCES:
- [Derived] Fawzy M, Emad M, Mahran A, Sabry M, Fetih AN, Abdelghafar H, Rasheed S. Artificial oocyte activation with SrCl2 or calcimycin after ICSI improves clinical and embryological outcomes compared with ICSI alone: results of a randomized clinical trial. Hum Reprod. 2018 Sep 1;33(9):1636-1644. doi: 10.1093/humrep/dey258. PMID 30099496